CLINICAL TRIAL: NCT05369260
Title: The Effect of Different Stabilization Exercises Based on Telerehabilitation on Gait, Balance, Functionality and Depression in Individuals With Non-Specific Chronic Neck Pain
Brief Title: Effect of Stabilization Exercises in Individuals With Non-Specific Chronic Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hatice AYAN, Lecturer, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOA-5309
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: Chronic Non-Spesific Neck Pain; Telerehabilitation; Gait; Balance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical and scapular stabilization group (Experimental): In this arm cervical and scapular stabilization exercises will be applied based on the telerehabilitation method via videoconference for 8 weeks, one day a week , 45-60 minutes for each session.
  Interventions: Other: Telerehabilitation-based cervical and scapular stabilization exercises
- Cervical and core stabilization group (Experimental): In this arm cervical and core stabilization exercises will be applied based on the telerehabilitation method via videoconference for 8 weeks, one day a week , 45-60 minutes for each session.
  Interventions: Other: Telerehabilitation-based cervical and core stabilization exercises

INTERVENTIONS:
Other: Telerehabilitation-based cervical and scapular stabilization exercises — Telerehabilitation based cervical and scapular stabilization exercises will be applied via videoconference method for 8 weeks, one day a week , 45-60 minutes for each session.
  Arms: Cervical and scapular stabilization group
Other: Telerehabilitation-based cervical and core stabilization exercises — Telerehabilitation based cervical and core stabilization exercises will be applied via videoconference method for 8 weeks, one day a week , 45-60 minutes for each session.
  Arms: Cervical and core stabilization group

SUMMARY:
In this study, the effects of an 8-week telerehabilitation-based stabilization training in persons with chronic non-specific neck pain will be investigated.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of different telerehabilitation-based stabilization exercises on gait, balance, pain, functionality and depression in individuals with non-specific neck pain. The population of the study will consist of 40 individuals with chronic neck pain, who are followed up with the diagnosis of chronic non-specific neck pain in the Department of Neurosurgery of Dokuz Eylul University Faculty of Medicine. The socio-demographic characteristics of the participants will be recorded through mutual interviews, 'BTS G-Walk' device for walking, 'Biodex Balance' device for balance, Neck Disability Index for disability assessment, Visual Analog Scale (VAS) for pain severity, the Beck Depression Inventory will be used for depression. All participants will walk to the length of a 10 m walkway and back to the start point with the BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device to assess spatiotemporal gait parameters. Individuals will walk first in a normal walking pattern and then in a fast walking pattern. Biodex Stability System will be used for balance measurement. The exercises will be taught to the participants face-to-face once in the first session, within the framework of social distance and hygiene rules, and then they will have exercise sessions by mutual videoconference method via the Zoom program for 8 weeks. Patients will be randomly divided into two groups. Cervical stabilization and scapular stabilization training will be given to the first group, and cervical stabilization and core stabilization training will be given to the second group. The effects of these two different telerehabilitation-based exercise methods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Having non-specific neck pain for at least 3 months
* Having a Neck Disability Index (BDI) score of 10 and above,

Exclusion Criteria:

* Receiving physiotherapy for neck pain in the last 6 months
* Having speech and comprehension problems,
* Those who have undergone neck surgery
* Those with sensory loss
* Those diagnosed with orthopedic, neurological or vestibular disease
* Those with a history of trauma ( wiplash)
* Cases diagnosed with cancer, osteoporosis or treated will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Speed | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess gait speed (m/sec) during usual walking condition and fast walking condition through a Bluetooth®3.0 connection (G-Studio®software).
Cadence | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess cadence (steps/min) during the usual walking condition and fast walking condition through a Bluetooth®3.0 connection (G-Studio®software).
Stride length | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess stride length (m) during the usual walking condition and fast walking condition through a Bluetooth®3.0 connection (G-Studio®software).
Step lenght | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess step length (% stride length) during in usual walking condition and fast walking condition through a Bluetooth®3.0 connection (G-Studio®software).
Gait Symmetry | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess gait symmetry. Gait symmetry index of the right and left sides are obtained during walking. The score is calculated by the device as a percentage score out of 100. The higher score indicates more symmetrical gait.
Pelvic angles | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess pelvic movements (tilt (°), obliquity(°), rotation(°)) during gait through a Bluetooth®3.0 connection (G-Studio®software). The device provides the data for these pelvic angles in one single report.
Pelvic symmetry | Change from Baseline at 8 weeks
  The BTS G-Walk (BTS Bioengineering S.p.A., GarbagnateMilanese, Italy), a wearable sensor device, will be used to assess pelvic symmetry (%) during gait through a Bluetooth®3.0 connection (G-Studio®software). The score is calculated by the device as a percentage score out of 100. The higher score indicates more pelvic symmetry.
Postural stability | Change from Baseline at 8 weeks
  A computerized test of the Biodex Balance System will be used to assess postural stability. Subjects will stand on the platform and try to maintain their stability while trying to control their center of pressure which is shown as a point on the screen. The postural stability test assesses the patient's ability to control static balance on a stable platform. The test protocol is performed for 20 seconds with 3 trials. The mean value of the trials is taken as a score. Higher stability index score indicates poor balance and stability.
Limits of stability | Change from Baseline at 8 weeks
  A computerized test of limits of stability will be performed using Biodex Balance System®. Subjects will stand on a stable platform and try to maintain their balance while trying to reach in different directions spot that is shown on the screen. The test results present scores for all directions. Higher scores show better performance (0= worst performance; 100= perfect performance).

SECONDARY OUTCOMES:
Neck Disability Index | Change from Baseline at 8 weeks
  Neck Disability Index will be used to evaluate the effects of neck pain on functional disability.
Visual Analog Scale (VAS) | Change from Baseline at 8 weeks
  It consists of a 10 cm horizontal or vertically positioned line on the page. The number '0', which is the starting point on this line, represents the patient's no pain, and the number '10' represents the worst pain experienced by the patient.
Beck Depression Inventory | Change from Baseline at 8 weeks
  It is designed to measure the severity of depression, to assess changes with treatment, and to identify the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Ayan, MSc, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- School of Physical Therapy and Rehabilitation, Dokuz Eylül University, Izmir, Turkey (Türkiye)